CLINICAL TRIAL: NCT05864638
Title: Acute Ischemic Stroke EndoVascular Therapy: a Multicenter REGISTRY Study （OCIN-AIS-EVT REGISTRY）
Brief Title: Acute Ischemic Stroke EndoVascular Therapy: a Multicenter REGISTRY Study
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jian-min Liu, Director of Cerebrovascular Disease Center, Changhai Hospital
Other Study IDs: OCIN-AIS-EVT REGISTRY
Record Dates: First submitted 2023-04-13; First posted 2023-05-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Thrombectomy; Thrombosis
MeSH Terms: conditions — Ischemic Stroke; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — thrombus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endovascular treatment
  Interventions: Device: Endovascular treatment

INTERVENTIONS:
Device: Endovascular treatment — Endovascular treatment, such as mechanical thrombectomy with stent, aspiration catheter or stent assisted by intermediate aspiration catheter, as well as combination of mechanical thrombectomy with intra-arterial thrombolysis

SUMMARY:
A Multicenter Registry of Endovascular Treatment for Acute Ischemic Stroke.

DETAILED DESCRIPTION:
The OCIN-AIS-EVT REGISTRY is a prospective, multicenter, blinded outcome evaluation, observational trial, and aims to determine the functional outcomes and safety of endovascular treatment for AIS, due to vessel occlusion in anterior and posterior circulation, in routine clinical practice.

The primary endpoint is functional outcome, defined as a shift (improvement) in scores on the modified Rankin scale (mRS) at 90 days (±7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke caused by anterior or posterior circulation vessel occlusion confirmed by computed tomography angiography (CTA) or magnetic resonance angiography (MRA) or digital subtraction angiography (DSA)
2. Undergo intravascular therapy (i.e. access to a cath lab and an arterial puncture)
3. The patient or his/her legal representative agreed to participate in the study and has signed the informed consent.

Exclusion Criteria:

1) No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All acute ischemic stroke patients receiving endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 90days
  Shift (improvement) in scores on the modified Rankin scale (mRS) at 90 days (±7 days). The value range 0-6: higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Dichotomized modified Rankin scale (mRS) | 90days
  Dichotomized modified Rankin scale (mRS) at 90 days after the procedure (0-1 versus 2-6, 0-2 versus 3-6, 0-3 versus 4-6). The value range 0-6: higher scores mean a worse outcome.
NIHSS at 24 hours | 24 hours post-procedure
  National Institutes of Health Stroke Scale (NIHSS) score at 24 hours post- procedure. The value range 0-42: higher scores mean a worse outcome.
NIHSS at 7 days | 7 days post procedure
  National Institutes of Health Stroke Scale (NIHSS) score at 7 days post procedure. The value range 0-42: higher scores mean a worse outcome.
Reperfusion outcome | Immediately post-procedure
  Immediate target vessel recanalization rate post-procedure: defined as proportion of subjects with extended thrombolysis in cerebral infarction (eTICI) score is 2b to 3 The value range 0-3: higher scores mean a better outcome.
Early successful revascularization rate | During procedure
  Early successful revascularization rate of target vessels by bridging therapy
Target vessel recanalization rate | at 7 days post-procedure
  Target vessel recanalization rate at 7 days post-procedure (assessed by CTA or MRA or DSA)

OTHER OUTCOMES:
Death | 7 days and 90 days
  All-cause death
Intracerebral hemorrhage(ICH) | 90 days
  Intracranial hemorrhage, including symptomatic intracranial hemorrhage (sICH) and asymptomatic intracranial hemorrhage
Procedure related complication | within 30 days after procedure
  Procedure related complication
Device related complications | within 30 days after procedure
  Device related complications
adverse events of special interest | within 90 days
  Other adverse events of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Jianimin Liu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Jianimin Liu, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses
URL: http://www.ocin.org.cn/about